CLINICAL TRIAL: NCT04124055
Title: Saliva and Dried Blood Spot Therapeutic Drug Monitoring for MDR-TB in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jan-Willem C Alffenaar (Other)
Collaborators: Kibong'oto Infectious Diseases Hospital (Other Government); University of Virginia (Other)
Responsible Party: Sponsor-Investigator, Jan-Willem C Alffenaar, prof, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-DBS-TDM-001
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: MDR-TB
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Drug Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapeutic drug monitoring (TDM) (Experimental): Therapeutic drug monitoring (TDM) based on Saliva and Dried blood spot samples
  Interventions: Diagnostic Test: Therapeutic drug monitoring (TDM)

INTERVENTIONS:
Diagnostic Test: Therapeutic drug monitoring (TDM) — Saliva and dried blood spot samples are collected. Based on the measured drug concentration the dose can be adjusted

SUMMARY:
Dried blood spot and saliva samples are collected during multidrug resistant tuberculosis (MDR-TB) treatment to measure the drug concentration of levofloxacin. Feasibility of both analytical procedures in a high burdened setting is explored.

DETAILED DESCRIPTION:
Background:

Measuring pharmacokinetic variability of anti-tuberculosis (TB) drugs and responding by dose correction will allow individualized treatment to improve microbiological response, curb acquired drug-resistance, protect and extend the efficacy of novel drugs rolled-out to endemic areas (pharmacovigilance), reduce toxicity to patients and lead to treatment duration shortening.

Aims and Objectives:

Implement Dried Blood Spot (DBS) collection for performance of high-performance liquid chromatography (HPLC) to optimize multidrug resistant TB (MDR-TB) treatment in Tanzania. Simultaneously, provide a proof-of-principle-demonstration that the developed saliva point of care drug assay for measurement of fluoroquinolone concentration works in a field setting.

Methods:

This will be a phase II prospective diagnostic study among patients from a national referral of MDR-TB in Tanzania. The investigators anticipate recruiting a minimum of 50 study participants to power for the primary aim. Subjects will have a minimum amount of blood and saliva collected for therapeutic drug monitoring and the investigational drug assays respectively. Expected results include agreement of saliva point-of-care and DBS for measurement of fluoroquinolone concentrations in HPLC. Other important findings related to field-testing include the best time for sample collection within the dosing interval and the algorithmic use of DBS and saliva, and clinical - demographic factors such as HIV coinfection, concomitant drugs, and diabetes mellitus that may influence the saliva drug assay results. Performance characteristics (sensitivity, specificity, negative and positive predictive values) of the saliva point-of care (PoC) and DBS will be calculated as a measurement of accuracy with reference to the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Participant is receiving care at Kibong'oto hospital
* Age of 18 years or above

Exclusion Criteria:

* Pregnancy at any gestation
* Co-morbid conditions such as generalized severe ulcers, Kaposi sarcoma,
* Hemophilia
* Participants with medical conditions like malignancy, dementia or those who will be critically ill and unable to consent and provide DBS and Saliva.
* Patients with Karnofsky score less than 40% or moribund

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Drug exposure | >2 weeks on treatment
  Drug concentration (mgL)

CONTACTS AND LOCATIONS:
Overall Officials: Stellah Mpagama, PhD, Principal Investigator — Kibong'oto ID hospital
Locations (1):
- Kibong'oto infectious diseases hospital, Kibong'oto, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohamed S, Mvungi HC, Sariko M, Rao P, Mbelele P, Jongedijk EM, van Winkel CAJ, Touw DJ, Stroup S, Alffenaar JC, Mpagama S, Heysell SK. Levofloxacin pharmacokinetics in saliva as measured by a mobile microvolume UV spectrophotometer among people treated for rifampicin-resistant TB in Tanzania. J Antimicrob Chemother. 2021 May 12;76(6):1547-1552. doi: 10.1093/jac/dkab057. PMID 33675664